CLINICAL TRIAL: NCT00101127
Title: A Phase II Evaluation of Docetaxel (NSC #628503) and Gemcitabine (NSC #613327) Plus G-CSF in the Treatment of Recurrent or Advanced Leiomyosarcoma of the Uterus
Brief Title: Docetaxel, Gemcitabine, and Filgrastim (G-CSF) or Pegfilgrastim in Treating Patients With Advanced, Persistent, or Recurrent Uterine Leiomyosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Masking: None | Purpose: Treatment
Other Study IDs: GOG-0087L; CDR0000405892
Record Dates: First submitted 2005-01-07; First posted 2005-01-10 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Sarcoma
Keywords: recurrent uterine sarcoma; stage III uterine sarcoma; stage IV uterine sarcoma; uterine leiomyosarcoma
MeSH Terms: conditions — Sarcoma | interventions — Filgrastim; pegfilgrastim; Docetaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: filgrastim
Biological: pegfilgrastim
Drug: docetaxel
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel and gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Colony-stimulating factors, such as G-CSF and pegfilgrastim, may increase the number of immune cells found in bone marrow or peripheral blood and may help the immune system recover from the side effects of chemotherapy. Giving docetaxel and gemcitabine together with G-CSF or pegfilgrastim may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving docetaxel and gemcitabine together with G-CSF or pegfilgrastim works in treating patients with advanced, persistent, or recurrent uterine leiomyosarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity of docetaxel, gemcitabine, and filgrastim (G-CSF) or pegfilgrastim in patients with advanced, persistent, or recurrent uterine leiomyosarcoma.
* Determine the nature and degree of toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to prior pelvic radiotherapy (yes vs no).

Patients receive gemcitabine IV over 90 minutes on days 1 and 8 and docetaxel IV over 1 hour on day 8. Patients also receive filgrastim (G-CSF) subcutaneously (SC) on days 9-15 OR pegfilgrastim SC on day 9. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 12-43 patients will be accrued for this study within 12-28 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed uterine leiomyosarcoma

  * Advanced, persistent, or recurrent disease
  * Documented disease progression
* Measurable disease

  * At least 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
* At least 1 target lesion

  * Tumors within a previously irradiated field are considered nontarget lesions
* Ineligible for higher priority GOG protocols (i.e., any active phase III GOG protocol for the same patient population)

PATIENT CHARACTERISTICS:

Age

* Adult

Performance status

* GOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN

Renal

* Creatinine ≤ 1.5 times ULN

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No neuropathy (sensory or motor) > grade 1
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer
* No active infection requiring antibiotics
* No known hypersensitivity to E. coli-derived proteins

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior cytotoxic chemotherapy for the malignancy

Endocrine therapy

* At least 1 week since prior hormonal therapy for the malignancy
* Concurrent hormone replacement therapy allowed

Radiotherapy

* See Disease Characteristics
* Recovered from prior radiotherapy

Surgery

* Recovered from prior surgery

Other

* Recovered from all other prior therapy
* No prior cancer treatment that would preclude study treatment
* No concurrent amifostine or other protective agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-12; Primary Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Antitumor activity
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Martee L. Hensley, MD, Study Chair — Memorial Sloan Kettering Cancer Center; Gregory P. Sutton, MD — St. Vincent Gynecologic Oncology at St. Vincent Oncology Center
Locations (60):
- United States (60):
  - Kaiser Permanente Medical Center - Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Helen and Harry Gray Cancer Center at Hartford Hospital, Hartford, Connecticut
  - New Britain General Hospital, New Britain, Connecticut
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - MBCCOP-Medical College of Georgia Cancer Center, Augusta, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Woman's Hospital, Baton Rouge, Louisiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Methodist Cancer Center at Methodist Hospital - Omaha, Omaha, Nebraska
  - Fox Chase Virtua Health Cancer Program - Marlton, Marlton, New Jersey
  - UMDNJ University Hospital, Newark, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - New York Oncology Hematology, PC at Albany Regional Cancer Care, Albany, New York
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Stony Brook University Cancer Center, Stony Brook, New York
  - Hope A Women's Cancer Center, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Forsyth Regional Cancer Center at Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center at Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Lake/University Ireland Cancer Center, Mentor, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Cancer Care Associates - Midtown Tulsa, Tulsa, Oklahoma
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Drexel University College of Medicine - Center City Hahnemann Campus, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Women and Infants Hospital of Rhode Island, Providence, Rhode Island
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Baptist Centers for Cancer Care, Memphis, Tennessee
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin

REFERENCES:
- [Result] Hensley ML, Blessing JA, Mannel R, Rose PG. Fixed-dose rate gemcitabine plus docetaxel as first-line therapy for metastatic uterine leiomyosarcoma: a Gynecologic Oncology Group phase II trial. Gynecol Oncol. 2008 Jun;109(3):329-34. doi: 10.1016/j.ygyno.2008.03.010. PMID 18534250